CLINICAL TRIAL: NCT00591396
Title: A Phase I Trial of ZIO-101 in Solid Tumors: Protocol # SGL1002
Brief Title: A Phase I Trial of ZIO-101 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL1002
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
MeSH Terms: interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ZIO-101 (Darinaparsin)

INTERVENTIONS:
Drug: ZIO-101 (Darinaparsin) — Dose Escalation of ZIO-101 (Darinaparsin) given daily for five consecutive days to be repeated every 28 days for up to six months
  Other Names: ZIO-101

SUMMARY:
A Phase I Trial of ZIO-101 (Darinaparsin) in Solid Tumors

ELIGIBILITY:
Inclusion Criteria

1. Subjects with histological confirmation solid malignancy refractory to conventional standard therapies for their condition
2. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions MUST not have been in a previously irradiated field or injected with biological agents
3. Pediatric subjects will be eligible at the discretion of the primary investigator.
4. ECOG performance status score ≤ 2
5. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative blood or urine pregnancy test within 1 week before beginning treatment. Sexually active men must also use acceptable contraceptive methods
6. Subjects must provide written informed consent prior to treatment
7. At least 4 weeks from prior completion of prior therapy to day 1 of study drug
8. Baseline toxicity assessment ≤ grade 1 except treatment induced alopecia (NCI Common Toxicity Criteria version 3.0)
9. Evidence of adequate multi-organ functional status as reflected by the following clinical laboratory values:

   * Serum creatinine ≤ 2 times the upper normal limit OR a calculated creatinine clearance ≥ 50 cc/min
   * Total bilirubin ≤ 2 times the upper normal limit
   * Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
10. Granulocytes in peripheral blood greater than or equal to 1 x 10(9) per liter, hemoglobin greater than or equal to 8.5 g/dL, and platelets greater than or equal to 50,000 /microL

Exclusion Criteria

1. Uncontrolled systemic infection (documented with microbiological studies)
2. Active heart disease as defined by an acute myocardial infarction within the previous 6 months before starting therapy, stable or unstable angina, clinically significant arrhythmia requiring medical management, OR New York Heart Association Classification of Functional Activities. Class 3: Subject has marked limitation in activities due to symptoms, even during less-than-ordinary activity and is comfortable only at rest OR Class 4: Severe limitations. Subject experiences symptoms even while at rest
3. Concomitant therapy for solid cancer
4. Pregnant subjects and those who are breast-feeding
5. History of an invasive second primary malignancy diagnosed within the previous 3 years except for Stage I Endometrial/Cervical Carcinoma or Prostate Carcinoma treated surgically, and non-melanoma skin cancer
6. Documented personal or family history of prolonged QT syndrome
7. 12 lead electrocardiogram with a corrected QT interval > 460 milliseconds
8. History of confusion or dementia
9. History of seizure disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States